CLINICAL TRIAL: NCT05549674
Title: The Copenhagen Cohort of Patients With Shoulder Pain: A Study Investigating Subacromial Impingement and Related Clinical Entities
Brief Title: Copenhagen Cohort of Patients With Shoulder Pain
Acronym: COPAIN
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Adam Witten, Medical Doctor, PhD student, Hvidovre University Hospital
Other Study IDs: COPAIN study
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Subacromial Impingement Syndrome; Subacromial Pain Syndrome; Subacromial Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The COPAIN study is observational. There is no intervention. — The COPAIN study is observational. There is no intervention.

SUMMARY:
The COPAIN study is comprised of three studies; a cross-sectional study (study 1), a prospective study (study 2) and a randomized controlled trial (study 3). Study 3 is described in detail in a separate protocol (the SELECT trial protocol) and is not described in further detail here.

DETAILED DESCRIPTION:
1. Study design

   Patients presenting with subacromial impingement syndrome (SIS) are subcategorized into clinical entities (section 6), including the entity 'isolated SI'. The distribution of patients within the different clinical entities is explored in study 1. Patients presenting with an entity other than isolated SI are treated in accordance with the preference of the treating shoulder surgeon. There is no formal follow-up of these patients within this project.

   Patients with isolated SI are prescribed at least three months of structured physiotherapy, and the correlation between the treatment outcome and individual pathophysiological factors (section 4) are investigated (study 2). Patients who does not benefit satisfactorily from at least 3 months of structured physiotherapy and presents with prolonged symptoms (at least 6 months) are offered to participate in a randomized controlled trial investigating the difference in treatment outcome from glenohumeral arthroscopy and ASD compared to glenohumeral arthroscopy alone (study 3). All patients are diagnosed and treated by orthopedic shoulder surgeons.
2. Research questions and objectives

   Study 1 1.31 Research question 1: Do patients with SIS constitute a heterogeneous group?

   Objective 1:

   To investigate how patients with SIS are distributed within predefined clinical entities.

   Study 2 Research question 2: Can individual pathophysiological factors predict the outcome after non-surgical treatment in patients with isolated subacromial impingement?

   Objective 2-A:

   To investigate if patients with a hook-shaped acromion have poorer outcome after non-surgical treatment than patients without a hook-shaped acromion.

   Objective 2-B:

   To investigate if patients with isolated SI and a positive scapular assistance test have better outcome from non-surgical treatment than patients without a positive scapular assistance test

   Objective 2-C:

   To investigate if other individual patient-related factors are correlated to the outcome after non-surgical treatment in patients with isolated SI.

   Study 3 (described in detail in the SELECT trial protocol) Research question 3: Is glenohumeral arthroscopy and arthroscopic subacromial decompression more effective than glenohumeral arthroscopy alone in improving patient-reported outcome in patients with isolated SI?
3. Outcomes

   Study 1 Outcome for objective 1 (To investigate how patients with SIS are distributed within clinical entities): The distribution of patients at baseline for each of the following entities; isolated subacromial impingement, full thickness rotator cuff tears, biceps tendinopathy, SLAP lesion, acromioclavicular osteoarthritis, minor shoulder instability and major shoulder instability.

   Study 2 Outcome for objective 2-A (To investigate if patients with isolated SI, that have a hook-shaped acromion, have poorer outcome from non-surgical treatment than patients without a hook-shaped acromion). The change in the Shoulder Pain and Disability Index (SPADI) 3 months after treatment was commenced.

   Outcome for objective 2-B (To investigate if patients with isolated SI, that have a positive scapular assistance test, have better outcome from non-surgical treatment than patients without a positive scapular assistance test). The change in the Shoulder Pain and Disability Index (SPADI) 3, 6 and 12 months after treatment was commenced.

   Outcome for objective 2-C (To investigate if other individual patient-related factors (section 5) are correlated to the outcome after non-surgical treatment in patients with isolated SI.) The change in the Shoulder Pain and Disability Index (SPADI) 3, 6 and 12 months after treatment was commenced.

   Study 3 Described in detail in the SELECT trial protocol.
4. Individual pathophysiological factors

   Acromial morphology

   Scapular assistance test The patients is asked to elevate the arm in the scapular plane as many degrees as possible while rating the level of shoulder pain using NPRS. The patient is then asked to elevate the arm again, but with the examiner manually facilitating the normal scapular movement. The test is considered positive if the patient reports less pain or is able to elevate the arm at least 10 degrees more when assisted by the examiner.
5. Other individual patient-related factors

   The following factors will be investigated for a possible association with the primary and secondary outcomes.

   Mechanical subacromial impingement The presence of mechanical subacromial impingement is examined with ultrasound and rated into one of the following categories: 1) not present, 2) present, but not consistently / only minor signs of mechanical impingement or 3) obviously present. This categorization is based on the findings from an unpublished pilot study. The participant is instructed to slowly elevate the arm in the scapular plane to 60 degrees while internally rotating 90 degrees. Mechanical impingement is defined as soft tissue impinging between the acromion and the humeral head.

   Scapular dyskinesis Scapula Dyskinesis is evaluated using the Scapula Dyskinesis Test (SDT). The SDT is a dynamic test in which the patient performs five repetitions of shoulder abduction and five repetitions of shoulder flexion while the rater observes for winging of the scapula and dysrhythmia. The SDT is rated as either obvious dyskinesis, slight dyskinesis or no dyskinesis.

   Critical shoulder angle (CSA) CSA is a radiological measurement of the angle between the glenoid inclination and the lateral border of the acromion.

   Subacromial bursa thickness and supraspinatus tendon thickness The bursa and tendon thickness are measured with ultrasound. The participant is asked to place the palm of the hand on the waist, with the elbow in 90 degrees flexion and directed lateral. The insertion of the supraspinatus tendon is visualized in the coronal plane. The thickness of both structures is measured 20 mm from the insertion of the supraspinatus tendon perpendicular to the tendon fibers.

   Acromio-humeral distance (AHD) The distance between the acromion and the humerus is measured with ultrasound. The participant is asked to keep the shoulder in neutral position with the arm relaxed. Acromion is visualized in the coronal plane and the AHD is measured as the shortest distance between the inferior edge of acromion and the upper edge of humerus.

   Subacromial injection test 5-10 ml lidocaine (10 mg/ml), with or without 40 mg corticosteroid, is injected into the subacromial space. Just before the injection the patient is asked to perform the shoulder movement provoking the most shoulder pain. After 5 minutes the patient is instructed to perform the same movement. The test is considered positive if the patient reports reduced shoulder pain.

   Background characteristics
   * Age (years)
   * Gender (male/female)
   * Dominant side affected (yes/no)
   * Shoulder demanding work/recreational activity (light physical demands / moderate demands / high demands)
   * BMI
   * Tobacco use (yes/no. If yes; pack-years)
   * Employment status (Employment status at the time of inclusion in the study (full time, part-time due to shoulder problems, part-time due to other reasons than shoulder problems, unemployed due to shoulder problems, unemployed due to other reasons than shoulder problems, sick leave due to shoulder problems, sick leave due to other reasons than shoulder problems, retired)
   * Marital status
   * Duration of symptoms (months)
6. Clinical entities

Rotator cuff tear Rotator cuff tears are diagnosed with ultrasonography or MRI. Tears are differentiated to be either partial thickness, full thickness or complete (partial thickness tears of the supraspinatus tendon is not considered a specific entity). A partial thickness tear is defined as a lesion that does not involve the whole thickness of the tendon. A full thickness tear extends through the whole thickness of the tendon, but not consistently. A complete tear is when the tendon has no connection to the footprint on the humerus.

Biceps tendinopathy The diagnosis is based on a clinical examination with findings of point tenderness in the bicipital groove and a positive Speed's test.

SLAP lesion A SLAP lesion is defined as an injury of the superior labrum of the glenohumeral joint. For the present study the diagnosis is synthesized from a positive O'Briens test and a typical patient history (repetitive overhead activity). Patients with an acute SLAP injury (not insidious onset of shoulder pain) are not included.

Acromioclavicular osteoarthritis Osteoarthritis of the acromioclavicular joint is defined as a positive cross-over test, recognizable pain at the acromioclavicular joint at palpation, and radiological signs of acromioclavicular osteoarthritis.

Shoulder instability Shoulder instability is divided into two clinical entities; minor shoulder instability and major shoulder instability. History of prior glenohumeral subluxations and/or dislocations are registered but is not determining for the clinical entity. Shoulder laxity is evaluated with the Sulcus test and the Load and shift test but does not alter the clinical entity. There is no time limit regarding previous glenohumeral subluxations/dislocations, but patients presenting with shoulder pain directly associated to a subluxation/dislocation (not insidious onset of shoulder pain), are not included.

1. Minor shoulder instability Pain from the Apprehension test or Castagna's test, but no signs of major instability.
2. Major shoulder instability 'Anterior instability' is defined as a positive Jobe´s apprehension test or Surprise test, and a positive Relocation test. 'Posterior instability' is defined as a positive jerk test.

ELIGIBILITY:
∙ At least 3 out of 5 positive tests from the following: Hawkin's test, Neer's test, Jobe's test, painful arc and external resistance test.

Insidious onset of pain

Exclusion criteria

* Terminal illness or severe medical illness (ASA score higher than or equal to 4)
* Systemic musculoskeletal disease
* Inflammatory joint disease (e.g. rheumatoid arthritis)
* Symptomatic cervical spine pathology
* Thoracic outlet syndrome
* Frozen shoulder
* Osteoarthritis of the glenohumeral joint
* Previous surgery, fracture or radiotherapy in the affected shoulder region
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with SIS referred to the place of investigation.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) 3 months after treatment is commenced. | 3 months
  SPADI is a patient-reported outcome measure designed to evaluate shoulder pain and disability. It ranges from 0 (best) to 100 (worst). It has 5 pain items and 8 disability items. The Danish version of SPADI has been found to have good reliability.

SECONDARY OUTCOMES:
Oxford Shoulder Score | Baseline, 3, 6 and 12 months
  Oxford Shoulder Score (OSS) is a patient-reported outcome measure specifically developed for assessing outcome after shoulder surgery. It ranges from 0 to 48, with 48 being the best. It contains 8 shoulder function items and 4 pain items, with each item scored from 0 to 4. It is validated in Danish and able to show change over time, with a Minimal Clinically Important Change (MCIC) of 6 points
EQ-5D-3L | Baseline, 3, 6 and 12 months
  EQ-5D-3L is a standardized patient-reported measure of health-related quality of life. It is a two-part instrument comprised of a descriptive system and a visual analogue scale (VAS). The descriptive system covers five dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression, that are each scored on a 3-level scale; no problems, some problems, and extreme problems. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number reflecting preferability compared to other health profiles. The VAS records the patient's self-rated health on a visual analogue scale with endpoints labelled 'Best imaginable health state and 'Worst imaginable health state'. This information can be used to compute quality-adjusted life years, which can be used in a cost-utility analysis to compare the benefit and cost of health care interventions.
Active shoulder abduction range of motion (AROM) | Baseline, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Witten A, Clausen MB, Thorborg K, Holmich P, Barfod KW. The Challenge of Diagnosing Patients Presenting With Signs and Symptoms of Subacromial Pain Syndrome: A Descriptive Study of 741 Patients Seen in a Secondary Care Setting. Orthop J Sports Med. 2025 Apr 28;13(4):23259671251332942. doi: 10.1177/23259671251332942. eCollection 2025 Apr. PMID 40303319